CLINICAL TRIAL: NCT01123070
Title: A Phase Ib Study Evaluating Safety, Pharmacokinetic and Pharmacodynamic Profiles of a Single Course of TL011 Infusions in Subjects With Severe, Active Rheumatoid Arthritis
Brief Title: TL011 in Severe, Active Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RA-TL011-101; 2009-015702-18 (EudraCT Number)
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TL011 (Experimental): TL011 infusions
  Interventions: Biological: TL011, anti CD20, for the treatment of rheumatoid arthritis
- MabThera (Active Comparator): MabThera infusions
  Interventions: Biological: MabThera infusions

INTERVENTIONS:
Biological: TL011, anti CD20, for the treatment of rheumatoid arthritis — TL011 administered by 2 infusions, 2 weeks apart
  Arms: TL011
Biological: MabThera infusions — MabThera, administered by 2 infusions, 2 weeks apart
  Arms: MabThera

SUMMARY:
The purpose of this study is to determine the safety and pharmacology of TL011 in patients with severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects
* Rheumatoid arthritis as defined by the 1987 ACR Classification
* Severe active seropositive disease
* Inadequate response or intolerance to other DMARDs
* Treatment with MTX

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* Active infection
* Known immunodeficiency syndrome
* Positive Hepatitis B surface antigen or antibodies to Hepatitis C
* History of cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-02-05 (Actual); Primary Completion 2012-04-23 (Actual); Study Completion 2012-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Czechia (3):
  - Teva Investigational Site 5428, Pilsen
  - Teva Investigational Site 5426, Prague
  - Teva Investigational Site 5429, Uherské Hradiště
- Hungary (4):
  - Teva Investigational Site 5123, Budapest
  - Teva Investigational Site 5122, Budapest
  - Teva Investigational Site 5125, Debrecen
  - Teva Investigational Site 5124, Szeged
- Italy (4):
  - Teva Investigational Site 3077, Florence
  - Teva Investigational Site 3075, Genova
  - Teva Investigational Site 3078, Pavia
  - Teva Investigational Site 3076, Siena
- Spain (4):
  - Teva Investigational Site 3170, Barakaldo
  - Teva Investigational Site 3168, Guadalajara
  - Teva Investigational Site 3167, Madrid
  - Teva Investigational Site 3169, Seville
- United Kingdom (3):
  - Teva Investigational Site 3434, Manchester
  - Teva Investigational Site 3433, Staffordshire
  - Teva Investigational Site 3435, Wirral, Merseyside

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A was an open label dose escalation for TL011 with two cohorts. Part B was randomized, double blind with two treatment groups to compare TL011 to MabThera. There was an 8 weeks core study period followed by 16 weeks extended follow up period.
Groups:
- Cohort 1 TL011 500 mg: Participants were administered 500 mg of TL011, via intravenous (IV) infusion, two weeks apart (on Day 1 and on Day 15).
- Cohort 2 TL011 1000 mg; Double Blind TL011 1000 mg: Participants were administered 1000 mg of TL011, via intravenous (IV) infusion, two weeks apart (on Day 1 and on Day 15).
- Double Blind MabThera 1000 mg: Participants were administered 1000 mg of MabThera, via intravenous (IV) infusion, two weeks apart (on Day 1 and on Day 15).
Period: Part A Cohort 1 Open Label Period
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Started | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A Cohort 2 Open Label Period
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Started | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part B Double Blind Period
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Started | 0 | 0 | 25 | 23
Completed | 0 | 0 | 21 | 20
Not Completed | 0 | 0 | 4 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Sponsor's Decision | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included participants that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg | Total
Number analyzed (Participants) | 3 | 3 | 25 | 23 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.56 (13.4) | 55.2 (8.3) | 56.8 (11.4) | 56.7 (12.2) | 56.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 22 | 18 | 45
  Male | 0 | 1 | 3 | 5 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Race : White | 3 | 3 | 24 | 23 | 53
  Race : Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve [AUC(0-t)] in Part B
Time Frame: Day 1 to Day 57
Population: Pharmacokinetics (PK) population included all participants that received at least one dose of 1000 mg TL011 or MabThera and had sufficient plasma concentration results to allow estimation of PK parameters
Measure: Geometric Mean (Standard Deviation); unit: Day*micrograms per milliliter
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 21 | 18
Day*micrograms per milliliter | 7571 (2219) | 8377 (2879)
Statistical Analysis 1: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; Test type: Equivalence — Bioequivalence declared if the back transformed 90% CI of geometric mean ratio is within the predefined limits of 0.75 to 1.33; p = 0.4265, ANCOVA; PK parameters were calculated using a logarithmic transformation. Covariates included body weight at screening, gender and treatment; Geometric mean ratio = 0.930, 90% CI 2-sided [0.797 to 1.084] — TL011 arm is the numerator and MabThera arm is the denominator

2. Secondary Outcome: Maximum Observed Concentration (Cmax) in Part B
Time Frame: Day 1 to Day 57
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 21 | 19
Micrograms per milliliter | 396 (84.2) | 450 (109)
Statistical Analysis 1: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0368, ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.862, 90% CI 2-sided [0.768 to 0.968] — TL011 arm is the numerator, MabThera arm is the denominator

3. Secondary Outcome: Number of Participants With Adverse Events in Part B
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as AEs occurring after the first dose of the study drug until 120 days after the last dose of study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From randomization up to Week 24
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 25 | 23
Participants | 14 | 16

4. Secondary Outcome: Cmax Post First Dose (C1max) and Post Second Dose (C2max) in Part B
Time Frame: Day 1, Day 15
Population: Pharmacokinetics (PK) population included all participants that received at least one dose of 1000 mg TL011 or MabThera and had sufficient plasma concentration results to allow estimation of PK parameters. Here, "number analyzed" signifies participants evaluable for this outcome measure. Numbers analyzed were not equal at each time point (C1max and C2max).
Measure: Geometric Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 22 | 22
Micrograms per milliliter
  C1max | 339 (68.2) | 356 (74.7)
  C2max: number analyzed (Participants) | 21 | 19
  C2max | 348 (124) | 448 (110)
Statistical Analysis 1: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; Cmax1; Test type: Equivalence — Bioequivalence declared if the 90% CI of geometric mean ratio is within the predefined limits of 0.75 to 1.33; p = 0.1484, ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.909, 90% CI 2-sided [0.814 to 1.014] — TL011/MabThera
Statistical Analysis 2: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; Cmax2; Test type: Equivalence — Bioequivalence declared if the 90% CI of geometric mean ratio is within the predefined limits of 0.75 to 1.33; p = 0.0241, ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.766, 90% CI 2-sided [0.633 to 0.927] — TL011/MabThera

5. Secondary Outcome: AUC At First Dose (AUC1) and AUC At Second Dose (AUC2) in Part B
Time Frame: Day 1, Day 15
Population: Pharmacokinetics (PK) population included all participants that received at least one dose of 1000 mg TL011 or MabThera and had sufficient plasma concentration results to allow estimation of PK parameters. Here, "number analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: Day*micrograms per milliliter
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 22 | 22
Day*micrograms per milliliter
  AUC1: number analyzed (Participants) | 20 | 19
  AUC1 | 2335 (527) | 2359 (634)
  AUC2: number analyzed (Participants) | 20 | 19
  AUC2 | 6133 (2774) | 6849 (4532)
Statistical Analysis 1: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; AUC1; Test type: Equivalence — Bioequivalence declared if the 90% CI of geometric mean ratio is within the predefined limits of 0.75 to 1.33; p = 0.6520, ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.969, 90% CI 2-sided [0.863 to 1.088] — TL011 arm is the numerator, MabThera arm is the denominator
Statistical Analysis 2: Comparison: Double Blind TL011 1000 mg vs Double Blind MabThera 1000 mg; AUC2; Test type: Equivalence — Bioequivalence declared if the 90% CI of geometric mean ratio is within the predefined limits of 0.75 to 1.33; p = 0.7835, ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.961, 90% CI 2-sided [0.757 to 1.222] — TL011/MabThera

6. Secondary Outcome: Percent Change From Baseline in CD19+ B-cell Count in Part B
Time Frame: Baseline to Day 57
Population: PK population. Here, "number analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 20 | 18
Percent change | -88.9 (25.9) | -90.6 (23.1)

7. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR20) Criteria Response in Part B
Description: Defined as at least 20% improvement from the screening values in swollen and tender joint count and in 3 of the following 5 disease activity measures.
  * Physician's global assessment of disease activity (VAS)
  * Patient's assessment of RA pain (VAS)
  * Patient's global assessment of disease activity
  * Patient's assessment of physical function (Health Assessment Questionnaire)
  * Acute phase reactant (C-reactive protein [CRP])
Time Frame: Baseline to Day 57
Population: Intent to Treat (ITT) population included all randomized participants regardless of the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
Number analyzed (Participants) | 25 | 23
Participants | 14 | 15

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve [AUC (0-t)] for Part A Cohort 2
Description: Data available for cohort 2 only per planned analysis.
Time Frame: Day 1 to Day 57
Population: Pharmacokinetics (PK) population included all participants that received at least one dose of 1000 mg TL011 and had sufficient plasma concentration results to allow estimation of PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: Day*micrograms per milliliter
Arm/Group | Cohort 2 TL011 1000 mg
Number analyzed (Participants) | 3
Day*micrograms per milliliter | 6423 (1956)

9. Secondary Outcome: Number of Participants With Adverse Events in Part A
Description: as for outcome 3
Time Frame: From randomization up to Week 24
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg
Number analyzed (Participants) | 3 | 3
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 24 weeks after first dose of study drug.
Description: Safety analysis set included all participants that received at least one dose of study treatment.
Arm/Group | Cohort 1 TL011 500 mg | Cohort 2 TL011 1000 mg | Double Blind TL011 1000 mg | Double Blind MabThera 1000 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/25 | 1/23
Other Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 11/25 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 TL011 500 mg (N=3) | Cohort 2 TL011 1000 mg (N=3) | Double Blind TL011 1000 mg (N=25) | Double Blind MabThera 1000 mg (N=23)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sideroblastic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 TL011 500 mg (N=3) | Cohort 2 TL011 1000 mg (N=3) | Double Blind TL011 1000 mg (N=25) | Double Blind MabThera 1000 mg (N=23)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.